CLINICAL TRIAL: NCT06101082
Title: An Exploratory Clinical Study Evaluating the Safety and Efficacy of Anti-HER2-CAR-T Cells Injection in Patients With HER2+ Locally Advanced and/ or Metastatic Solid Tumors
Brief Title: A Clinical Study Evaluating the Safety and Efficacy of Anti-HER2-CAR-T Cells Injection in Patients With Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: China Medical University, China (Other)
Collaborators: Shanghai First Song Therapeutics Co., Ltd (Industry)
Responsible Party: Principal Investigator, Funan Liu, professor, China Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HER2-CN-A1
Record Dates: First submitted 2023-10-20; First posted 2023-10-25 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Solid Tumor
Keywords: CAR-T; solid tumor; Cell therapy; HER2
MeSH Terms: interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-HER2-CAR-T cell infusion (Experimental): Anti-HER2-CAR-T cell is administered as a single intravenous infusion. Follow-up infusions are based on the investigator's decision.The dose group to be infusion was 1×10^6 CAR-T cells/kg, 3×10^6 CAR-T cells/kg, and 1×10^7 CAR-T cells/kg based on the 3+3 dose escalation principle. The infusion dose refers to the number of CAR-positive cells.The patients will receive lymphocyte clearance therapy with cyclophosphamide and fludarabine before the infusion.
  Interventions: Biological: Intravenous infusion anti-HER2-CAR-T cell

INTERVENTIONS:
Biological: Intravenous infusion anti-HER2-CAR-T cell — Anti-HER2-CAR-T cell is administered as a single intravenous infusion. Follow-up infusions are based on the investigator's decision.The dose group to be infusion was 1×10^6 CAR-T cells/kg, 3×10^6 CAR-T cells/kg, and 1×10^7 CAR-T cells/kg based on the 3+3 dose escalation principle. The infusion dose refers to the number of CAR-positive cells.
  Other Names: fludarabine; cyclophosphamide

SUMMARY:
This is a single-center, open-label clinical study of anti-HER2-CAR-T cells for HER2+ patients with locally advanced and/or metastatic solid tumors. In this study, a single-dose regimen was designed, and the investigator had the discretion to decide whether the patient received more than once CAR T-cell therapy.This study intends to include HER2+ patients with locally advanced and/or metastatic solid tumors.They will take the anti-HER2-CAR-T cell transfusion after a screening period, mononuclear cell (PBMC) collection, bridging therapy if necessary, and lymphocyte clearance pretreatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients should understand and sign informed consent forms and voluntarily participate in clinical studies;
2. Age≥ 18, < 70 years old, gender is not limited;
3. Locally advanced and/or metastatic solid tumors; HER2-positive expression in tumor tissues (staining 3+, or staining 2+ with HER2 gene amplification should be further performed by ISH and other methods) ;
4. Histology-confirmed solid tumors (breast cancer,gastric cancer, colorectal cancer, pancreas cancer, etc.), conventional treatment is ineffective or Intolerability conventional treatment or lack of effective treatment;
5. According to RECIST v 1.1, at least one measurable lesion with a maximum lesion diameter not exceeding 6 cm;
6. Expected survival≥ 12 weeks;
7. ECOG score≤ 2 ;
8. Adequate hematological function ; have no performed blood transfusion or received cell growth factor within 7 days before screening hematological evaluation:Neutrophil ≥ 1.0×10^9/L;Hemoglobin≥ 80g/L;Platelet ≥ 75×10^9/L;Lymphocytes ≥ 0.5×10^9/L
9. Adequate liver function: serum total bilirubin ≤1.5× ULN (excluding Gilbert's syndrome); AST and ALT≤2.5×ULN( AST and ALT ≤5×ULN with liver metastasis);
10. Adequate renal function: creatinine ≤1.5× ULN or endogenous creatinine clearance ≥50 mL/min;
11. LVEF ≥ 50%;
12. There was no evidence that subjects had difficulty breathing at rest or pulse oximetry>90% when breathing indoor air;
13. Sufficient intravenous access for apheresis; no other contraindications to blood cell separation;
14. The pregnancy test for women of childbearing age must be negative. All subjects must agree to take effective contraception from the signing of the informed consent to 6 months after the last dose of the study drug infusion.

Exclusion Criteria:

1. Previously using any CAR-T cell products or other genetically modified T cell therapies;
2. Patients who are waiting for organ transplantation or with a history of allogeneic stem cell or solid organ transplantation;
3. Patients with acute or uncontrolled active infection, including but not limited to active tuberculosis;
4. Patients with Hepatitis B infection (HBV surface antigen positive and/or hepatitis B core antibody positive and hepatitis B DNA >10^3 copies /mL) ; hepatitis C infection(hepatitis C antibodies positive) ; Syphilis infection (antibody positive), HIV infection (antibody positive);
5. Patients with hyponatremia and/or hypokalemia, blood sodium <125mmol/L and/or blood potassium<3.5mmol/L (Sodium and/or potassium supplementation may be given before participating in the study to restore blood sodium and/or potassium above this level);
6. Imaging results the proportion of liver replaced by tumor ≥50%;
7. Patients who taken continuous systemic steroids within 14 days before apheresis or within 72 hours before cell therapy (prednisone> 5 mg/day or equivalent dose of other hormones), excepting for those who use inhaled Steroid hormones;
8. Systemic sexualization is accepted 2 weeks before apheresis or 5 half-lives (whichever is shorter). Toxicity to previous antineoplastic therapy has not recovered (based on CTCAE version 5.0 assessment); excepting for alopecia, pigmentation and other tolerable events judged by the investigator or permitted laboratory 9.abnormalities according to the protocol;
9. Antibody therapy within 4 weeks before apheresis and preconditioning;
10. Anti-PD-1/PD-L1 monoclonal antibody therapy within 4 weeks before apheresis and preconditioning;
11. Immunostimulation or immunosuppressive therapy within 28 days prior to apheresis;
12. Radiotherapy within 28 days prior to apheresis, except limited local palliative radiotherapy;
13. Patients with other malignant tumors within the past 5 years or at the present (except for basal cell carcinoma of the skin, breast/cervix Carcinoma in situ and other malignant tumors that have not been treated in the past five years have been effectively controlled);
14. Patients with active ulcers or active gastrointestinal bleeding that are difficult to control;
15. Patients with previous medical history of central nervous system (CNS) primary or metastatic tumors including meningeal metastases, unless previously treated for brain metastases, who are currently asymptomatic, and do not need steroid or enzyme-inducing antiepileptic drug treatment within 14 days before screening;
16. Patients with other central nervous system diseases that may affect the safety of the subjects as judged by the researchers (such as epileptic seizures, cerebral hemorrhage, dementia, etc.);
17. Patients with uncontrolled hypertension, unstable angina, NYHA III or higher-grade congestive heart failure with an ejection fraction of the heart below 50%, or an ECG with significant abnormalities, serious arrhythmias requiring treatment and medical history of myocardial infarction within 6 months prior to initiation of study treatment;
18. Patients with severe respiratory diseases before apheresis, such as interstitial lung disease, active pulmonary tuberculosis;
19. Patients with active or past autoimmune diseases that may relapse (such as systemic lupus erythematosus, rheumatoid arthritis, etc.), except for the following diseases: type 1 diabetes, hypothyroidism that only needs hormone replacement therapy, skin diseases that do not require systemic therapy (such as vitiligo, psoriasis or hair loss);
20. Any serious or uncontrollable systemic disease, systemic Complications, other serious concurrent diseases (such as hemophagocytic syndrome, etc.), special cases of tumor conditions according to the investigator's judgment that may make patients unsuitable for entry into the study or affect compliance with the protocol, or significant interference with the correct assessment of drug safety, toxicity, and effectiveness;
21. Received any major surgery within 4 weeks before apheresis (except exploratory laparotomy or laparoscopy exploration) or severe trauma; Any major surgery during the DLT observation period, or has not yet completely recovered from any previous invasive procedure;
22. Patient allergic or intolerant to the preconditioning drugs that may be used in the research process or the drugs for symptomatic treatment of CRS , including but not limited to fludarabine and cyclophosphamide or tocilizumab;Known hypersensitivity to the components of anti-HER2-CAR-T; or have any history of severe allergies, for example, anaphylactic shock;
23. Patients who have participated in other interventional clinical trials within 1 month before administration;
24. Pregnant or lactating women;
25. Patients of childbearing age who are unwilling or unable to use reliable contraception during the study period;
26. Patients who are unable or unwilling to comply with clinical protocols as judged by the investigator;
27. Persons involved in the study plan and execution.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2026-10-19 (Estimated); Study Completion 2026-10-19 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity | 21 days within anti-HER2-CAR-T cell infusion
  Dose-limiting toxicity

SECONDARY OUTCOMES:
Objective response rate | 4week,8week,3month,6month,9month and12month after the anti-HER2-CAR-T cell infusion
  Objective response rate

CONTACTS AND LOCATIONS:
Overall Officials: Zhenning Wang, doctor, Principal Investigator — The First Affiliated Hospital of China Medical Univeristy; Funan Liu, doctor, Principal Investigator — The First Affiliated Hospital of China Medical Univeristy
Locations (1):
- Phase I Clinical Trials Center Of The First Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No